CLINICAL TRIAL: NCT02627768
Title: Assessment of STELARA® (Ustekinumab) and Tumor Necrosis Factor Alpha Inhibitor Therapies in Patients With Psoriatic Arthritis in Standard Health-Care Practice; A Prospective, Observational Cohort
Brief Title: A Study on Assessment of STELARA and Tumor Necrosis Factor Alpha Inhibitor Therapies in Participants With Psoriatic Arthritis
Acronym: PsaBio
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106450; CNTO1275PSA4003 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Psoriatic Arthritis
Keywords: STELARA; Psoriatic Arthritis; Ustekinumab
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Ustekinumab Treatment: Participants who have a confirmed diagnosis of Psoriatic Arthritis (PsA) and are starting ustekinumab as a first, second, or third line of biological disease-modifying antirheumatic drugs (bDMARD) therapy.
  Interventions: Drug: No Intervention
- Cohort 2: TNFi Treatment: Participants who have a confirmed diagnosis of Psoriatic Arthritis (PsA) and are starting a tumor necrosis factor alpha inhibitor (TNFi) as a first, second, or third line of biological disease-modifying antirheumatic drugs (bDMARD) therapy.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — Participants who have a confirmed diagnosis of Psoriatic Arthritis (PsA) and are starting ustekinumab or a tumor necrosis factor alpha inhibitor (TNFi) as a first, second, or third line of biological disease-modifying antirheumatic drugs (bDMARD) therapy will be observed.

SUMMARY:
The purpose of this study is to evaluate treatment retention in psoriatic arthritis participants with STELARA or tumor necrosis factor alpha inhibitor (TNFi) therapies in relation to effectiveness, safety, benefit/risk and to examine clinical response.

DETAILED DESCRIPTION:
This is a prospective, observational, cohort study to collect data on adult participants who have a confirmed diagnosis of psoriatic arthritis (PsA) and are starting either STELARA or a new TNFi as a new therapy in a first, second, or third line of biologic disease-modifying antirheumatic drug (bDMARD) therapy. Approximately 1,400 participants will be enrolled into this study, with 700 participants who are receiving STELARA at study entry and 700 participants who are receiving a new TNFi therapy at study entry. Recruitment into the study will continue for approximately 2 years (with the possibility to extend this period if the patient enrollment target is not reached), with a 3-year follow-up period. For each participant, the follow-up period will continue for 3 years (36 months) after inclusion into the study. Participants will primarily be assessed for parameters of treatment retention, clinical response, effectiveness and safety over an observational period of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of psoriatic arthritis (PsA) as determined by a rheumatologist according to ClASsification criteria for Psoriatic Arthritis (CASPAR) criteria
* Must be starting either STELARA or any new approved tumor necrosis factor alpha inhibitor (TNFi) (including TNFi biosimilar) as a new biologic disease-modifying antirheumatic drug (bDMARD) therapy in a first, second or third line of bDMARD therapy for PsA at the time of enrollment into the observational study or within a maximum 2-month window after the baseline visit
* Must sign a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Participant is starting STELARA or a TNFi therapy as fourth or further line of biologic treatment
* Participant is unwilling or unable to participate in long-term data collection
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before the start of the study or the first data collection time point
* Participant is currently enrolled in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have a confirmed diagnosis of Psoriatic Arthritis (PsA) and are starting either STELARA or a new tumor necrosis factor alpha inhibitor (TNFi) as a new therapy in a first, second, or third line of biological disease-modifying antirheumatic drugs (bDMARD) therapy.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Time to Drug Stop or Switch | Up to Month 36
  Time taken to stop or switch the study drug is evaluated.
Change From Baseline in Disease Activity Score in 28 Joints (DAS28) at Month 36 | Baseline and Month 36
  The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: 0 = no disease activity to 100 = maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. European League Against Rheumatism (EULAR) Good response: DAS28 less than or equal to (<=) 3.2 or a change from Baseline less than (<) -1.2. EULAR Moderate response: DAS28 greater than (>) 3.2 to <= 5.1 or a change from Baseline < -0.6 to greater than or equal to (>=) -1.2.
Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) Scores at Month 36 | Baseline and Month 36
  The DAPSA score will be calculated by the data collection tool and is the sum of the following: Participant's assessment of pain on visual analog scale (VAS) (in centimeters), Participant's Global Assessment of Disease Activity on VAS, 66 and 68 joint counts for swelling and tenderness, respectively. Joints assessed include the distal interphalangeal (DIP), proximal interphalangeal (PIP), and metacarpophalangeal (MCP) joints of the hands; the wrist, elbow, shoulder, acromioclavicular, sternoclavicular, temporomandibular, hip (excluded for swelling), knee, ankle, and midtarsal joints; and the metatarsophalangeal and PIP joints of the feet. CRP level in milligrams per deciliters (mg/dL). Cut-off values for low and high disease activity are <= 14 and > 28 points, respectively, and for remission is <= 4 points.
Percentage of Participants Achieving Low Disease Activity Based on DAPSA Score | Month 36
  The DAPSA score will be calculated by the data collection tool and is the sum of the following: Participant's assessment of pain on VAS (in centimeters), Participant's Global Assessment of Disease Activity on VAS, 66 and 68 joint counts for swelling and tenderness, respectively. Cut-off values for low and high disease activity are <= 14 and > 28 points, respectively, and for remission is <= 4 points.
Percentage of Participants Achieving Remission Based on DAPSA Score | Month 36
  The DAPSA score will be calculated by the data collection tool and is the sum of the following: Participant's assessment of pain on VAS (in centimeters), Participant's Global Assessment of Disease Activity on VAS, 66 and 68 joint counts for swelling and tenderness, respectively. Cut-off values for low and high disease activity are <= 14 and > 28 points, respectively, and for remission is <= 4 points.
Change From Baseline in Physician's Global Assessment of Disease Activity (PGA-PsA) Measured on a Visual Analogue Scale at Month 36 | Baseline and Month 36
  Physician's and Patient's Global Assessment of Disease Activity (PGA) are measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity).
Change From Baseline in Patient Global Assessment of Disease Activity (PtGA) at Month 36 | Baseline and Month 36
  The PtGA VAS is a self-administered assessment with scores ranging from "very well" (0 mm) to "very poor" (100 mm) that assesses disease activity over the past week. Proposed categories for interpretation of the VAS score: <10 mm, low disease activity; >= 10 millimeter (mm) but <30 mm moderate disease activity; >= 30 mm but <60 mm high disease activity; >= 60 mm very high disease activity.
Percentage of Participants with Dactylitis Over Time | Up to Month 36
  The total number of digits of the hands and feet (that is, 0 to 20) with dactylitis will be evaluated.
Percentage of Participants with Enthesitis Over Time | Up to Month 36
  Enthesitis will be documented using the Leeds Enthesitis Index (LEI). The LEI examination points include the lateral epicondyle (left and right), medial femoral condyle (left and right), and Achilles tendon insertion (left and right).
Change From Baseline in Nail Involvement Scores (Number Of Nails) at Month 36 | Baseline and Month 36
  Nail involvement will be evaluated by recording the total number of nails of the hands and feet (that is, 0 to 20) with PsA involvement.
Change From Baseline in C-Reactive Protein (CRP) at Month 36 | Baseline and Month 36
  C-Reactive Protein will be evaluated to measure the inflammation.
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Month 36 | Baseline and Month 36
  Erythrocyte Sedimentation Rate will be evaluated to measure the inflammation.
Percentage of Participants With Body Surface Area (BSA) Psoriasis (PsO) Skin Involvement | Month 36
  Psoriasis skin involvement will be documented using categories: <3 percentage (%), 3% to 10%, and >10% of BSA. The typical method to assess BSA is to consider the surface area of the participant's handprint (palm and fingers) as representing 1% of the body's surface area.
Change From Baseline in Body Surface Area (BSA) Psoriasis (PsO) Skin Involvement at Month 36 | Baseline and Month 36
  Psoriasis skin involvement will be documented using categories: <3%, 3% to 10%, and >10% of BSA. The typical method to assess BSA is to consider the surface area of the participant's handprint (palm and fingers) as representing 1% of the body's surface area.
Percentage Change From Baseline in EuroQoL 5-Dimension 3-Level Questionnaire (EQ-5D-3L) Scores at Month 36 | Baseline and Month 36
  The EQ-5D-3L is a standardized measure of health status developed by the EuroQoL Group to provide a simple, generic measure of health for clinical and economic appraisal. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical economic evaluation of health care. The EQ 5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, severe problems.
Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Month 36 | Baseline and Month 36
  The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a participant completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A participant must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Percentage of Participants Achieving in the Health Assessment Questionnaire Disability Index (HAQ-DI) Response | Month 36
  The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a participant completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A participant must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Change From Baseline in Psoriatic Arthritis Impact of Disease-12 (PsAID-12) at Month 36 | Baseline and Month 36
  The PsAID-12 is a validated, self-administered questionnaire developed by EULAR for use in clinical practice that assesses the impact of PsA on participants' lives. It consists of 12 questions, each answered using a numerical rating scale. Questions related to pain, skin problems, work and/or leisure activities, discomfort, embarrassment and/or shame, social participation, and anger, fear, and uncertainty; and depression are scored from 0 (none) to 10 (extreme), functional capacity and sleep disturbance are scored from 0 (no difficulty) and 10 (extreme difficulty) and coping is scored from 0 (very well) 10 (very poorly).
Change From Baseline in Pain Visual Analogue Scale (VAS) Scores at Month 36 | Baseline and Month 36
  The pain VAS is a self-administered assessment of average pain during the past week. The scale ranges from "no pain" (0 mm) to "the worst possible pain" (100 mm). This assessment should be completed prior to the tender and swollen joint examination.
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Scores at Month 36 | Baseline and Month 36
  The BASDAI participant rated components over last 48 hours using 100 mm Visual Analog Scale; components 15: range 0=none to 100=very severe; component 6: range:0=0 hours to 100=2 hours or more. 1) Overall level of fatigue/tiredness experienced; 2) Overall level of AS neck,back or hip pain experienced; 3) Overall level of pain/swelling in joints other than neck, back or hips; 4) Overall level of discomfort from any areas tender to touch or pressure; 5) Overall level of morning stiffness from time of awakening; 6) Duration of morning stiffness from time of awakening, and morning stiffness sub-scale.
Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Psoriatic Arthritis (WPAI:PsA) Scores at Month 36 | Baseline and Month 36
  The WPAI:PsA is a validated, self-administered questionnaire that assesses work and activity impairment during the past 7 days. The WPAI:PsA produces 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on the job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI: PsA outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Percentage of Participants With Change in Employment Status | Month 36
  Change in the employment status of participants will be evaluated.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (Approximately Month 39)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (66):
- Belgium (9):
  - Brussels
  - Céroux-Mousty
  - Forest
  - Genk
  - Gilly
  - Hasselt
  - Leuven
  - Liège
  - Merksem
- France (12):
  - Besançon
  - Bordeaux
  - Clermont-Ferrand
  - Corbeil
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Montpellier, Herault
  - Paris
  - Toulouse
  - Tours
- Greece (6):
  - Athens
  - Heraklion
  - Larissa
  - Pátrai
  - Thessaloniki
  - Voula Attica
- Netherlands (7):
  - Alkmaar
  - Amsterdam
  - Den Helder
  - Groningen
  - Rotterdam
  - Sneek
  - Utrecht
- Russia (6):
  - Kemerovo
  - Khabarovsk
  - Moscow
  - Saint Petersburg
  - Saransk
  - Stavropol
- Spain (10):
  - Barcelona
  - Bilbao
  - Donostia / San Sebastian
  - Getafe
  - Granada
  - Madrid
  - Mérida
  - Salamanca
  - Valladolid
  - Vitoria-Gasteiz
- United Kingdom (16):
  - Abergavenny
  - Bath
  - Cambridge
  - Cannock
  - Christchurch
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Reading
  - Salford
  - Sheffield
  - Stoke-on-Trent
  - Wigan
  - Wolverhampton

REFERENCES:
- [Derived] Alle G, Lopez-Medina C, Siebert S, Lavie F, Noel W, Smolen JS, Gossec L. Patient Profiles in Randomized Controlled Trials Versus a Real-World Study in Psoriatic Arthritis: Scoping Review and Metaanalysis. J Rheumatol. 2025 Feb 1;52(2):138-144. doi: 10.3899/jrheum.2024-0653. PMID 39547694
- [Derived] Gossec L, Siebert S, Bergmans P, de Vlam K, Gremese E, Joven-Ibanez B, Korotaeva TV, Lavie F, Noel W, Nurmohamed MT, Sfikakis PP, Sharaf M, Theander E, Smolen JS. Improvement in patient-reported outcomes and work productivity following 3-year ustekinumab or tumour necrosis factor inhibitor treatment in patients with psoriatic arthritis: results from the PsABio real-world study. Arthritis Res Ther. 2023 Jun 23;25(1):109. doi: 10.1186/s13075-023-03058-y. PMID 37353788
- [Derived] Van Kuijk AWR, Nurmohamed MT, Siebert S, Bergmans P, de Vlam K, Gremese E, Joven-Ibanez B, Korotaeva TV, Lavie F, Sharaf M, Noel W, Theander E, Smolen JS, Gossec L, van der Horst-Bruinsma IE. Gender-specific differences in patients with psoriatic arthritis receiving ustekinumab or tumour necrosis factor inhibitor: real-world data. Rheumatology (Oxford). 2023 Oct 3;62(10):3382-3390. doi: 10.1093/rheumatology/kead089. PMID 36810788
- [Derived] Gossec L, Siebert S, Bergmans P, de Vlam K, Gremese E, Joven-Ibanez B, Korotaeva TV, Lavie F, Noel W, Nurmohamed MT, Sfikakis PP, Sharaf M, Theander E, Smolen JS. Long-term effectiveness and persistence of ustekinumab and TNF inhibitors in patients with psoriatic arthritis: final 3-year results from the PsABio real-world study. Ann Rheum Dis. 2023 Apr;82(4):496-506. doi: 10.1136/ard-2022-222879. Epub 2022 Dec 13. PMID 36600178
- [Derived] Gossec L, Siebert S, Bergmans P, de Vlam K, Gremese E, Joven-Ibanez B, Korotaeva TV, Lavie F, Noel W, Nurmohamed MT, Sfikakis PP, Theander E, Smolen JS. Persistence and effectiveness of the IL-12/23 pathway inhibitor ustekinumab or tumour necrosis factor inhibitor treatment in patients with psoriatic arthritis: 1-year results from the real-world PsABio Study. Ann Rheum Dis. 2022 Jun;81(6):823-830. doi: 10.1136/annrheumdis-2021-221640. Epub 2022 Feb 24. PMID 35210262